CLINICAL TRIAL: NCT05450653
Title: Pilot Trial of Fetoscopic Endoluminal Tracheal Occlusion (FETO) in Fetuses With Severe Congenital Diaphragmatic Hernia (CDH)
Brief Title: Trial of FETO for Severe Congenital Diaphragmatic Hernia
Acronym: FETO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aimen F. Shaaban, MD (Other)
Responsible Party: Sponsor-Investigator, Aimen F. Shaaban, MD, Director, Chicago Institute for Fetal Health, Principal Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Organization: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-4085
Record Dates: First submitted 2022-06-14; First posted 2022-07-11 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: Hernia, Diaphragmatic, Congenital; Fetal Endoscopic Tracheal Occlusion; Fetoscopic Endoluminal Tracheal Occlusion; Pregnant; Humans; Fetoscopy
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Hernia, Diaphragmatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- FETO with GOLDBAL2 (Experimental): A detachable balloon will be inserted in the fetal airway during the FETO procedure.
  Interventions: Device: FETO with Goldballoon Detachable Balloon (GOLDBAL2) along with the delivery Microcatheter (BALTACCI-BDPE100)

INTERVENTIONS:
Device: FETO with Goldballoon Detachable Balloon (GOLDBAL2) along with the delivery Microcatheter (BALTACCI-BDPE100) — A Goldballoon Detachable Balloon (GOLDBAL2) will be inserted in the airway of the fetus with severe congenital diaphragmatic hernia (o/e LHR <25% with liver up) during the FETO procedure between gestational age 27 weeks 0 days and 29 weeks and 6 days. The fetal tracheal balloon will be removed at between 34 weeks 0 days and 34 weeks 6 days gestation or earlier as indicated.

SUMMARY:
This is a single site pilot trial to study the feasibility of Fetoscopic Endoluminal Tracheal Occlusion (FETO) therapy in the most severe group of fetuses with congenital diaphragmatic hernia (CDH) at Ann & Robert H. Lurie Children's Hospital of Chicago (Lurie Children's). This procedure aims to increase fetal lung volume before birth and improve survival after birth. This study will enroll 10 pregnant women who meet study criteria.

DETAILED DESCRIPTION:
A Goldballoon Detachable Balloon (GOLDBAL2) will be inserted into the fetal trachea and deployed with the Delivery Microcatheter (BALTACCI-BDPE100) between 27 weeks 0 days and 29 weeks and 6 days of gestation. The fetal tracheal balloon will be removed between 34 weeks 0 days and 34 weeks 6 days of gestation or earlier as indicated.

After balloon insertion, participants will be followed weekly and must reside within 30 minutes of Lurie Children's until balloon removal. Additionally, participants will have restrictions from return to work, exercise, or intercourse. The children's health status will be followed until two years of age.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Pregnant individuals age 18 years and older
* Singleton pregnancy
* No pathogenic variants on prenatal chromosomal microarray or pathologic findings on karyotype analysis. Results by fluorescence in situ hybridization (FISH) will be acceptable if the patient is > 26 weeks
* Isolated left CDH with severe pulmonary hypoplasia with o/e LHR </=25% with liver up (measured at 18 weeks 0 days to 29 weeks 5 days of gestation) OR Isolated right CDH with severe pulmonary hypoplasia with o/e LHR </=35% with liver up (measured at 18 weeks 0 days to 29 weeks 5 days of gestation)
* Gestational age at FETO procedure 27 weeks 0 days to 29 weeks 6 days as determined by clinical information and evaluation of first ultrasound
* Fetal echocardiogram with changes expected with CDH and no major structural cardiac defects
* Stated willingness to comply with all study procedures and lifestyle considerations and availability for the duration of the study

  * Willingness to reside within 30 minutes of the Chicago Institute for Fetal Health (CIFH) in the time period between the FETO placement procedure and the balloon retrieval procedure and ability to maintain follow up appointments
  * Subject has a support person (e.g., spouse, partner, friend, parent) that is available to stay with her for the duration of the pregnancy near Lurie Children's
  * Willingness to comply with study restrictions on work, exercise, and intercourse
* Meets psychosocial criteria

Exclusion Criteria:

* Rubber latex allergy
* Presence of chromosomal abnormalities or anatomic anomalies that are known to significantly alter survival prognosis (i.e., CDH and congenital heart disease). No cases will be removed post hoc if abnormalities are discovered during post-operative monitoring
* History of preterm labor, cervix shortened to ≤20 mm at enrollment or at 24 hours prior to FETO balloon insertion procedure) or uterine anomaly strongly predisposing to preterm labor or placenta previa
* Maternal contraindication to fetoscopic surgery or severe maternal medical condition in pregnancy
* History of incompetent cervix with or without cerclage
* Placental abnormalities (previa, abruption, accreta, chorioangioma) known at time of enrollment
* Maternal-fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy
* Maternal HIV, Hepatitis-B, Hepatitis-C status positive because of the increased risk of transmission to the fetus during maternal-fetal surgery. If the patient's HIV or Hepatitis status is unknown, the patient must be tested and found to have negative results before enrollment
* Uterine anomaly such as large or multiple fibroids or mullerian duct abnormality
* There is no safe or technically feasible fetoscopic approach to balloon placement
* Participation in another intervention study that influences maternal and fetal morbidity and mortality
* Any other condition which, in the opinion of the investigator, would compromise safety, feasibility or impede compliance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-09-18 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Number of successful placements of Goldballoon Detachable Balloon at gestational age 27 weeks 0 days (27w0d) to 29 weeks 6 days (29w6d) | 27 weeks zero days to 29 weeks 6 days
  Successful completion of balloon insertion in fetuses with severe CDH defined as direct visualization of balloon above the carina at the time of FETO procedure.
Number of successful removals of balloon | Removal prior to delivery, ideally at 34 weeks gestation
  Removal of the balloon will ideally be done at 34th week of gestation or prior to delivery.

SECONDARY OUTCOMES:
Change in fetal lung growth | Baseline (before balloon placement) to first ultrasound after balloon removal
  Prenatal ultrasound will measure the observed-to-expected lung to head ratio (o/e LHR) at weekly visits while the balloon is in place and after balloon removal. Fetal lung growth will be calculated as the difference between the o/e LHR pre-balloon placement and the o/e LHR after balloon removal.
Gestational age at delivery | At the time of delivery
  Gestational age at delivery will be recorded.
Infant survival | Birth to 24 months
  Infant survival will be measured from delivery to discharge, at 6, 12, and 24 months of age.
Number of infants requiring extra corporeal membrane oxygenation (ECMO) support | Birth to 6 months
  Use of ECMO will be collected from medical chart review.
Number of infants with sepsis | Birth to six months
  Sepsis occurrences will be collected from medical chart review.
Number of infants with intraventricular hemorrhage (IVH) | Birth to six months
  Intraventricular hemorrhage data will be collected from medical chart review.
Length of hospital stay | Birth to one year
  Hospital length of stay will be calculated from medical chart review.
Number of infants requiring supplemental oxygen | Birth to 24 months
  Supplemental oxygen requirement at time of discharge will be collected from medical chart review.
Number of maternal complications | Up to 4-6 weeks post-partum
  Complications during pregnancy, delivery, and first post-partum visit to include: preterm labor, premature rupture of membranes (PROM), preterm premature rupture of membranes (PPROM), oligohydramnios, polyhydramnios, placental abruption, chorioamnionitis, and other infection.

CONTACTS AND LOCATIONS:
Overall Officials: Aimen Shaaban, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MedlinePlus Genetics: Congenital diaphragmatic hernia — https://medlineplus.gov/genetics/condition/congenital-diaphragmatic-hernia/
- See also: Genetic and rare diseases information resources: Congenital Diaphragmatic Hernia — https://rarediseases.info.nih.gov/diseases/1481/congenital-diaphragmatic-hernia
- See also: U.S. FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks
- See also: Hernia — https://medlineplus.gov/hernia.html